CLINICAL TRIAL: NCT00595010
Title: Developing Multi-Component Evidence Based Practice in Child Abuse Service Systems
Brief Title: Effectiveness of a Multi-Component Evidence-Based Parent Training Program in Reducing Child Maltreatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R34MH076972 (NIH); R34MH076972 (NIH)
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Child Abuse
Keywords: Child Maltreatment; Child Neglect; Child Physical Abuse; Evidence-Based Practice

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Managing Child Behavior (Experimental): Families with a high risk for or a history of child abuse and are enrolled in Comprehensive Home-Based Services and receive services as usual, which includes SafeCare, plus Managing Child Behavior module if they report significant behavior problems with their child between the ages of 2-12.
  Interventions: Behavioral: SafeCare

INTERVENTIONS:
Behavioral: SafeCare — Treatment will be based on an updated version of the SafeCare program, which specifically addresses parenting and discipline associated with child physical abuse. Participants will receive services from Comprehensive Home-Based Services.

SUMMARY:
This study will determine the effectiveness of a complex parent training program, based on the SafeCare model, in reducing the occurrence of child maltreatment.

DETAILED DESCRIPTION:
Child maltreatment is the general term used to characterize all forms of child abuse, including neglect and physical, sexual, and emotional abuse. These forms of maltreatment can lead to a large number of child developmental, emotional, and behavioral difficulties. As adults, children who are maltreated are more prone to unhealthy behaviors and conditions, such as drug and alcohol abuse, smoking, eating disorders, and depression. A previous study found that Project SafeCare, a treatment program that provides parent training to families with children who were at risk for or victims of maltreatment, resulted in fewer child welfare reports. Participants in Project SafeCare reported improvements in child healthcare, home safety, and parent-child relations. However, the study suggested that the SafeCare program may not be equally effective in decreasing the occurrence of all forms of child maltreatment, particularly child physical abuse. This study will determine the effectiveness of a complex evidence-based practice program, extending upon the SafeCare program, in reducing the occurrence of physical abuse and other forms of child maltreatment.

Participants in this study will receive services from Oklahoma Comprehensive Home-Based Services (CHBS), a program provided to families with issues of child abuse and neglect. Upon entry into the CHBS program, participants will undergo a computerized interview, lasting between 1 and 2 hours. The interview will include questions about family strengths and weaknesses, personal beliefs, substance abuse history, and opinion on CHBS. This computerized interview will be repeated at the end of treatment, approximately 6 to 12 months later. During the first few weeks of CHBS, an agent will make five visits to the homes of participants to observe pretreatment family life. Treatment services will concentrate on improving healthcare skills, parent-child interactions, and safety in homes and will specifically address ways to reduce physical abuse and other identified family issues. Study participation will continue for 12 months after completion of CHBS. Study researchers will obtain child welfare reports from the Department of Human Services (DHS) for up to 10 years after completion of CHBS.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Oklahoma Comprehensive Home-Based Services (CHBS)
* Child referred by Office of Community Services

Exclusion Criteria:

* Primary referral of sexual abuse
* Primary referral goal to maintain permanent placement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Fidelity of service provider | Measured throughout study

SECONDARY OUTCOMES:
Parent behavior | Measured at baseline and at some point between Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Debra B. Hecht, PhD, Principal Investigator — University of Oklahoma

IPD SHARING:
Plan to Share IPD: No